CLINICAL TRIAL: NCT00527566
Title: Mepolizumab As a Steroid Sparing Treatment Option in the Churg Strauss Syndrome
Brief Title: Mepolizumab As a Steroid-sparing Treatment Option in the Churg Strauss Syndrome
Acronym: MATOCSS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Michael Wechsler, MD, Assistant Professor of Medicine at Harvard Medical School and Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-P-000012/1;BWH
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Churg Strauss Syndrome
Keywords: Churg Strauss Syndrome
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mepolizumab (Experimental): Subjects will receive open-label mepolizumab
  Interventions: Biological: Mepolizumab

INTERVENTIONS:
Biological: Mepolizumab — IV mepolizumab, 750 mg
  Other Names: Anti IL-5

SUMMARY:
The purpose of this study is to determine whether Mepolizumab (a monoclonal antibody against interleukin-5) is a safe and well-tolerated therapy that will allow for steroid tapering in patients with steroid-dependent Churg-Strauss Syndrome (CSS).

DETAILED DESCRIPTION:
Specific Aims:

1. Document the safety of mepolizumab therapy in patients with CSS.
2. Demonstrate the steroid sparing effect of mepolizumab therapy by decreasing corticosteroid dosage while using this anti-IL5 therapy.
3. Demonstrate the efficacy of anti-IL5 therapy in improving the signs and symptoms of CSS by:

   1. Measuring serum markers of CSS disease activity, including: peripheral eosinophilia, erythrocyte sedimentation rate, anti- neutrophil cytoplasmic antigen, C-reactive protein and IgE levels.
   2. Assessing the activity level of vasculitis via the Birmingham Vasculitis Activity Score
   3. Evaluating asthmatic response via serial peak flow and FEV1 measurements as well as asthma symptom scores using the Juniper scale.
   4. Assessing changes in novel parameters such as fractional excretion of nitric oxide and IL-5 levels.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Diagnosis of Churg Strauss Syndrome
* Maintained on stable corticosteroid dose of at least prednisone 10mg daily (or equivalent) prior to enrollment in study
* If on cyclophosphamide, azathioprine or methotrexate, must be on a stable dose and be able to maintain that dose for the duration of the study

Exclusion Criteria:

* Hypereosinophilic Syndrome
* Wegener's Granulomatosis
* Malignancy
* Parasitic Disease
* Pregnant or nursing
* If female and of child-bearing potential, must have negative pregnancy test prior to each infusion of study medication and must adhere to acceptable method of contraception (with <1% failure rate)
* Any other medical illness that precludes study involvement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wechsler, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Martin RM, Wilton LV, Mann RD. Prevalence of Churg-Strauss syndrome, vasculitis, eosinophilia and associated conditions: retrospective analysis of 58 prescription-event monitoring cohort studies. Pharmacoepidemiol Drug Saf. 1999 May;8(3):179-89. doi: 10.1002/(SICI)1099-1557(199905/06)8:33.0.CO;2-K. PMID 15073927
- [Background] Harrold LR, Andrade SE, Go AS, Buist AS, Eisner M, Vollmer WM, Chan KA, Frazier EA, Weller PF, Wechsler ME, Yood RA, Davis KJ, Platt R. Incidence of Churg-Strauss syndrome in asthma drug users: a population-based perspective. J Rheumatol. 2005 Jun;32(6):1076-80. PMID 15940771
- [Background] Hellmich B, Csernok E, Gross WL. Proinflammatory cytokines and autoimmunity in Churg-Strauss syndrome. Ann N Y Acad Sci. 2005 Jun;1051:121-31. doi: 10.1196/annals.1361.053. PMID 16126951
- [Background] Garrett JK, Jameson SC, Thomson B, Collins MH, Wagoner LE, Freese DK, Beck LA, Boyce JA, Filipovich AH, Villanueva JM, Sutton SA, Assa'ad AH, Rothenberg ME. Anti-interleukin-5 (mepolizumab) therapy for hypereosinophilic syndromes. J Allergy Clin Immunol. 2004 Jan;113(1):115-9. doi: 10.1016/j.jaci.2003.10.049. Epub 2003 Dec 12. PMID 14699394
- [Background] Stein ML, Collins MH, Villanueva JM, Kushner JP, Putnam PE, Buckmeier BK, Filipovich AH, Assa'ad AH, Rothenberg ME. Anti-IL-5 (mepolizumab) therapy for eosinophilic esophagitis. J Allergy Clin Immunol. 2006 Dec;118(6):1312-9. doi: 10.1016/j.jaci.2006.09.007. Epub 2006 Nov 7. PMID 17157662
- [Background] Plotz SG, Simon HU, Darsow U, Simon D, Vassina E, Yousefi S, Hein R, Smith T, Behrendt H, Ring J. Use of an anti-interleukin-5 antibody in the hypereosinophilic syndrome with eosinophilic dermatitis. N Engl J Med. 2003 Dec 11;349(24):2334-9. doi: 10.1056/NEJMoa031261. No abstract available. PMID 14668459
- [Background] Menzies-Gow A, Flood-Page P, Sehmi R, Burman J, Hamid Q, Robinson DS, Kay AB, Denburg J. Anti-IL-5 (mepolizumab) therapy induces bone marrow eosinophil maturational arrest and decreases eosinophil progenitors in the bronchial mucosa of atopic asthmatics. J Allergy Clin Immunol. 2003 Apr;111(4):714-9. doi: 10.1067/mai.2003.1382. PMID 12704348
- Available data/document: Publication: PubMed ID: 20513524 — http://www.ncbi.nlm.nih.gov/pubmed/20513524 — Mepolizumab as a steroid-sparing treatment option in patients with Churg-Strauss syndrome. Kim S, Marigowda G, Oren E, Israel E, Wechsler ME. J Allergy Clin Immunol. 2010 Jun;125(6):1336-43. doi:10.1016/j.jaci.2010.03.028.

RESULTS

PARTICIPANT FLOW:
Groups:
- Mepolizumab: Intravenously infused 750 mg of mepolizumab 1x every 4 weeks for 16 weeks.
Period: Overall Study
Arm/Group | Mepolizumab
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Participants: # White Participants | 7
  Participants: Unknown | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Indicated Side Effects
Description: Side effects experienced by participants 1 to 2 days after Mepolizumab infusion.
Time Frame: Participants were followed for the duration of the study, approximately 44 weeks
Measure: Number; unit: Participants
Arm/Group | Mepolizumab
Number analyzed (Participants) | 10
Participants
  Mild transient headaches | 3
  Mild pruritus | 1
  Urticaria, allergic reaction, worsening symptoms | 0
  Loose stool | 1

2. Secondary Outcome: Steroid Dosing During Trial
Time Frame: 20 weeks
Measure: Mean (Full Range); unit: Prednisone mg/day
Arm/Group | Mepolizumab
Number analyzed (Participants) | 10
Prednisone mg/day
  Baseline (Week 0) | 14.3 [10 to 20]
  Week 12 | 5.6 [2 to 12.5]
  Week 20 | 4.9 [0 to 20]

3. Secondary Outcome: Evaluate Overall Positive Change in Churg-Strauss Syndrome Via the Measures Outlined in Study Aims
Description: The Asthma Control Questionnaire (ACQ) was one measure used to assess the prevalence of asthma symptoms the participant was having during the study. It is a series of 7 questions assessing how often, over the past two weeks, the participant wakes up from their asthma, how bad their symptoms were, etc. The greater the prevalence of symptoms, the higher the score. Each of the 7 questions is scored 0-6. The total score is calculated by adding the individual question scores and dividing the sum by 7.
Time Frame: 20 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Mepolizumab
Number analyzed (Participants) | 10
units on a scale
  Week 0, baseline | 1.40 [0 to 2.86]
  Week 12, Treatment phase | 1.76 [0.29 to 7]
  Week 20, end of washout phase | 1.30 [0 to 4.1]

4. Primary Outcome: Number of Participants Who Experienced Specific Symptoms
Description: Number of participants who experienced specific symptoms during the trial.
Time Frame: 44 weeks
Measure: Number; unit: Participants
Arm/Group | Mepolizumab
Number analyzed (Participants) | 10
Participants
  Wheeze or cough | 4
  Sore throat | 4
  Nausea or abdominal discomfort | 3
  Sinusitis | 6
  Arthritis | 1

5. Secondary Outcome: Efficacy- Exacerbation Rate
Description: Quantified the exacerbation rate (total number of exacerbations per day) of the participants during treatment with mepolizumab and without treatment. Exacerbations were characterized as any worsening of clinical disease requiring an increase of systemic corticosteroid therapy (e.g. prednisone) for asthma, respiratory symptoms, or underlying vasculitis.
Time Frame: Treatment period (12 weeks)
Measure: Number; unit: Exacerbation rate (Exacerbations/day)
Groups:
- Mepolizumab (Treatment Phase): Intravenously infused 750 mg of mepolizumab 1x every 4 weeks for 16 weeks.
- Non-treatment Phase: The non-treatment phase consists of the wash-out phase and the safety monitoring phase.
Arm/Group | Mepolizumab (Treatment Phase) | Non-treatment Phase
Number analyzed (Participants) | 10 | 10
Exacerbation rate (Exacerbations/day) | 0.14 | 0.69

ADVERSE EVENTS:
Arm/Group | Mepolizumab
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab (N=10)
Fractured Hip (Musculoskeletal and connective tissue disorders) | 1 (1) — Subject fell and broke hip. Event classified as serious, unexpected, and unrelated.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab (N=10)
Headache (Nervous system disorders) | 4 (5)
Digestive System Issues (Gastrointestinal disorders) | 3 (3) — Abdominal pain/diarrhea, gastroenteritis, gastroesophageal reflux
Churg-Strauss Syndrome Flair (Endocrine disorders) | 3 (5)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Wheezing and Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No